CLINICAL TRIAL: NCT01416766
Title: CONtrolling Disease Using Inexpensive IT - Hypertension in Diabetes
Acronym: CONDUIT-HID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Reliant Medical Group (Other); University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, Barry Saver, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CONDUIT-001; R18HS018461 (AHRQ)
Record Dates: First submitted 2011-08-03; First posted 2011-08-15 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Hypertension; Diabetes Mellitus
Keywords: Blood Pressure Monitors; Medical Informatics; Disease Management; Comparative Effectiveness Research
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Control participants will receive usual care during their year of enrollment. At enrollment, prior to randomization, they will be informed that, if randomized to control status, they will be offered a free BP monitor and the opportunity to receive the study intervention after completing the exit interview in 1 year.
- Intervention (Experimental): Self-monitoring-nurse-primary care provider feedback loop After randomization, intervention participants will receive the intervention (free home BP monitor, assistance setting up to upload BP readings from home/work or clinic computer; feedback loop with nurse-driven protocols to manage uncontrolled hypertension and maintain control once attained).
  Interventions: Other: Self-monitoring-nurse-primary care provider feedback loop

INTERVENTIONS:
Other: Self-monitoring-nurse-primary care provider feedback loop — Intervention participants will receive an Omron BP monitor and assistance in setting it up to upload BP data to Reliant Medical Group from a home/work or clinic-based computer. They will be encouraged to upload readings at least once/month. Diabetes management nurses will receive the readings and, if a participant's mean BP is not at target, will follow protocols to address this, contacting PCPs as indicated by protocols.
  Other Names: CONDUIT blood pressure intervention
  Arms: Intervention

SUMMARY:
This project will develop and test a low-cost approach to using health information technology and home monitoring aimed at improving care for chronic conditions, with low barriers to adoption in a wide variety of settings - from large group practices using state-of-the-art electronic health records to small practices with no more than a computer with internet access. Success will lead to a cost-effective approach to improving control of hypertension, both among individuals with diabetes and among non-diabetics, which can make a substantial contribution to the health of the population of the United States as improving hypertension control is estimated to have a greater population health benefit than most other health interventions. Success will also set the stage for adaptation of this intervention to a variety of other chronic health conditions and further substantial improvements in the health of millions of Americans.

DETAILED DESCRIPTION:
This project will develop and test a low-cost approach to using health information technology (HIT), aimed at improving the effectiveness and cost-effectiveness of care for chronic health conditions that are amenable to home self-monitoring, that is easy to disseminate. In contrast to many other HIT-based interventions, the investigators will utilize commercial, off-the-shelf technology rather than custom, expensive HIT. The investigators are using hypertension control among persons with diabetes as our test case because there is documented need for improving control of hypertension in this high-risk population and studies estimate that improving hypertension control in diabetes is more cost-effective than most other medical interventions and possibly even cost-saving in direct health care dollars. This high-value return on investment is important for encouraging adoption, expansion, and dissemination of HIT innovations. Our intervention will involve recruiting 400 persons with diabetes and uncontrolled hypertension receiving care through Reliant Medical Group (RMG - formerly called Fallon Clinic). MODIFICATION (2/13) - Due smaller than anticipated numbers of eligible persons and low enrollment, we are expanding eligibility to include "prediabetics". Half of them will be randomly assigned to receive an automated blood pressure (BP) monitor capable of uploading readings through a computer, plus instruction on how to connect their monitors at home or in the clinic to upload their information into a popular and free commercial personal health record (PHR) system. These blood pressure data from the PHR will be transferred automatically into RMG's electronic health record (EHR) system and will alert RMG's existing team of care management nurses. Subjects whose blood pressure is uncontrolled will have their medication regimens intensified by these nurses according to protocols. Intervention subjects will receive regular outreach calls from the care management nurses if their blood pressure remains uncontrolled or they are not periodically uploading blood pressure readings. After one year, the investigators will compare outcomes between control and intervention subjects. Our primary outcomes will be change in mean blood pressure and proportion of subjects with controlled blood pressure. The investigators will also measure a range of secondary outcomes including costs of the intervention, medication utilization, and a variety of patient-reported outcomes. Furthermore, the investigators will interview and observe study subjects and care providers to gain a better understanding of factors affecting uptake and use of the intervention. The investigators will examine continued use of the intervention after formal study participation ends and will also measure uptake of the intervention by control subjects offered delayed entry at the end of the formal study. Lastly, the investigators will compare our study and findings to other, recent studies using HIT to improve hypertension control and develop a set of best practices and recommendations for future efforts in this area.

ELIGIBILITY:
Inclusion Criteria:

* diagnoses of both diabetes mellitus (MODIFICATION 2/13: prediabetes) and hypertension
* uncontrolled hypertension (mean of up to most recent 3 clinic BPs in previous 6 months with SBP>=145 and/or DBP>=85) AND mean of 3 readings taken at intake visit meeting same criterion

Exclusion Criteria:

* end-stage renal disease
* management of blood pressure by provider other than primary care provider (PCP)
* pregnancy/gestational diabetes
* terminal illness
* diagnosed or probable (based on screen) dementia
* active psychosis
* moderate-severe mental retardation
* indication by PCP that patient would be inappropriate for study
* planning to leave Reliant Medical Group (formerly Fallon Clinic) during the coming year

MODIFICATIONS: due to a smaller pool of eligible participants and lower enrollment than anticipated, eligibility for the study has been expanded as of February 2013 to include persons with "prediabetes," defined by either a coded diagnosis of abnormal glucose (International Classification of Diseases [ICD] 9-CM codes 790.2x) or a hemoglobin A1c laboratory value from 6.0%-6.4%. For this group, the DBP eligibility criterion will be a mean, as defined above, of >=95, as target BP for this group is 140/90, not 140/80.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2011-08; Primary Completion 2014-10 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure (BP) | At entry (day 1) and 1 year later; secondarily, electronic health record (EHR)-based readings prior to entry and one year later
  We will assess differences in changes in systolic BP (SBP) and diastolic BP (DBP) measured at study intake and 1 year later at exit. We will also evaluate changes in mean EHR BP readings prior to study entry and in the 3 months before study exit. We will also assess the primary outcome in terms of % of intervention vs. control participants achieving control (originally proposed as mean of 3 exit readings <130 SBP and 80 DBP but now revised to 140 SBP and 80 DBP due to new evidence and change in the Healthcare Effectiveness Data and Information Set (HEDIS) measure for 2011). NOTE: For eligible participant group added 2/13, "prediabetic" patients, DBP control will be judged as mean <90mmHg as target BP for these groups is 140/90.

SECONDARY OUTCOMES:
Refill adherence | 6 months prior to study entry and 6 months prior to study exit
  We will compare changes in the Medication Possession Ratio for antihypertensive medications for the 6 months prior to study entry and the 6 months prior to study exit for the subset of participants for whom insurance claims give us complete data on prescription fills.
Self-reported medication adherence | At entry (day 1) and 1 year later, at exit
  Change in self-reported medication adherence, based on: 1) the modified Morisky scale and 2) a visual analog scale (Walsh).
Technology use | Continuous over course of study; final measurement at exit interview for intervention subjects & 6 mos. after exit for controls
  We will measure use of home/office/other personal computers to upload BP readings over the internet vs. bringing BP monitor to clinic and uploading data vs. calling/mailing/faxing readings (offered to those not doing either of the first 2 after 2-3 months). We intend to offer delayed entry after the exit to control subjects and will assess their use over the next 3-6 months.
Health care utilization | Enrollment through exit 1 year later
  We will measure counts of Reliant Medical Group visits and hospitalizations. Number of antihypertensive medications and post/pre change will be compared for control vs. intervention participants. We will also compare health care costs, as represented by billed charges; complete charges are expected to be available for ~70% of participants; clinic-only charges will be compared for the remainder.
Satisfaction | At entry (day 1) and 1 year later, at exit
  Participant satisfaction with care will be measured using Consumer Assessment of Healthcare Providers and Systems (CAHPS) clinician and group survey questions.

CONTACTS AND LOCATIONS:
Overall Officials: Barry G Saver, MD, MPH, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- Reliant Medical Group, Worcester, Massachusetts, United States

REFERENCES:
- [Result] Marquard JL, Garber L, Saver B, Amster B, Kelleher M, Preusse P. Overcoming challenges integrating patient-generated data into the clinical EHR: lessons from the CONtrolling Disease Using Inexpensive IT--Hypertension in Diabetes (CONDUIT-HID) Project. Int J Med Inform. 2013 Oct;82(10):903-10. doi: 10.1016/j.ijmedinf.2013.04.009. Epub 2013 Jun 22. PMID 23800678